CLINICAL TRIAL: NCT07047950
Title: The Effect of Health Belief Model-Based Education and Counseling Program on Coronary Heart Disease Risk
Brief Title: Effect of Health Belief Model-Based Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Muhammet Faruk Yigit, Assistant Professor Dr., Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ınonu university
Record Dates: First submitted 2025-04-21; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases Risk; Health Belief Model; Nursing
Keywords: Cardiovascular Diseases, Health Belief Model
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: A quasi-experimental design with a pre-test and post-test approach was employed.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No intervention applied
- Experimental group (Experimental): * Implementation of the HBM Based Individual Education and Counseling Program for the Prevention of CHD
  * Phone calls conducted in the 2nd and 4th months after education.
  * Educational booklet distributed
  Interventions: Behavioral: Individual Education and Counseling Program

INTERVENTIONS:
Behavioral: Individual Education and Counseling Program — The educational programme entitled "HBM Approach to Prevent CHD" was designed by the researcher and delivered as a presentation. The educational sessions were conducted face-to-face at the Cardiology Outpatient Clinic of Van Yüzüncü Yıl University Dursun Odabaş Medical Center and lasted approximately 35-45 minutes. In addition, follow-up telephone calls were made to individuals in the intervention group twice at two-month intervals.
  The content of the educational programme was developed based on a comprehensive literature review using resources from the Turkish Society of Cardiology, the WHO, the Ministry of Health, the Turkish Public Health Institution, evidence-based research and previous studies. The programme covered topics such as the definition of CHD, risk factors, treatment, complications, perceived susceptibility and severity of CHD, perceived benefits, barriers and strategies to overcome them, self-efficacy, and rules for engaging in physical activity and maintaining a health
  Arms: Experimental group

SUMMARY:
Aim: This study aimed to determine the impact of an education and counseling program based on the health belief model on coronary heart disease risk factors knowledge level, risk perception of heart disease, and Framingham risk scores.

Background: Coronary heart disease remains a leading cause of morbidity and mortality worldwide, and effective prevention strategies are critical. The health belief model provides a theoretical framework for understanding and influencing health behaviors. A quasi-experimental design with a pre-test and post-test approach was employed.

Methods: Data were collected using the Descriptive Characteristics Form, the Cardiovascular Disease Risk Factors Knowledge Level Scale, and the Heart Disease Risk Perception Scale. Additionally, Framingham risk scores were calculated.

DETAILED DESCRIPTION:
The educational programme entitled "HBM Approach to Prevent CHD" was designed by the researcher and delivered as a presentation. The educational sessions were conducted face-to-face at the Cardiology Outpatient Clinic of Van Yüzüncü Yıl University Dursun Odabaş Medical Center and lasted approximately 35-45 minutes. In addition, follow-up telephone calls were made to individuals in the intervention group twice at two-month intervals.

The content of the educational programme was developed based on a comprehensive literature review using resources from the Turkish Society of Cardiology, the WHO, the Ministry of Health, the Turkish Public Health Institution, evidence-based research and previous studies. The programme covered topics such as the definition of CHD, risk factors, treatment, complications, perceived susceptibility and severity of CHD, perceived benefits, barriers and strategies to overcome them, self-efficacy, and rules for engaging in physical activity and maintaining a healthy diet.

Participants in the educational sessions received a booklet entitled "Health Belief Model Approach to Prevent CHD" as a reminder tool. This booklet contained the same information as the presentation.

The education was given to the intervention group immediately after the collection of the pre-test data. The control group received no intervention. The post-test data were collected six months after the pre-test. After the post-test, participants in the control group also received the educational booklet.

The care approach, based on the HBM, included several interventions aimed at increasing participants' awareness of CHD. To increase the perception of susceptibility, participants were informed about the definition, symptoms, incidence and risk factors of CHD, thereby increasing their sensitivity to the issue. To increase perceptions of severity, the health, social and economic problems caused by CHD were explained in detail. Perceptions of benefits were enhanced by emphasising the benefits of prevention in the lives of the participants.

In terms of barriers, potential obstacles to adopting health-promoting behaviours to prevent CHD were explained in detail. Health motivation was supported by providing education and counselling services to help participants overcome these barriers. Finally, in the self-efficacy dimension, participants were encouraged to share their thoughts about prevention methods, which helped to build their confidence. This approach aimed to empower participants to be more aware and effective in preventing CHD.

ELIGIBILITY:
Inclusion Criteria:

* Being under the age of 65
* Having normal cognitive functioning
* Having no communication difficulties

Exclusion Criteria:

* Not volunteering to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Knowledge Level of Cardiovascular Disease Risk Factors Scale | From 01 January 2023 to 01 Februrary 2023 (4 weeks)
  The Knowledge Level of Cardiovascular Disease Risk Factors Scale (KL-CDRFS) was developed and validated by Arıkan et al. in 2009. Notably, it is the inaugural scale in Turkey to have been both validated and proven reliable for the purpose of assessing knowledge levels concerning cardiovascular disease risk factors (Cronbach's alpha: 0.768). The scale comprises 28 items, and evaluation is based on the total score obtained.
Demographic Information Form | From 01 January 2023 to 01 Februrary 2023 (4 weeks)
  The form comprises 17 questions with the objective of gathering information about patients' age, gender, education level, employment status, presence of chronic diseases, medication use, marital status, family history of heart disease, prior knowledge about heart diseases, information on prevention of heart diseases, smoking status, systolic blood pressure, diastolic blood pressure, HDL cholesterol, LDL cholesterol, fasting blood glucose levels, and Framingham risk scores.
Perception of Heart Disease Risk Scale | From 01 January 2023 to 01 Februrary 2023 (4 weeks)
  The Perception of Heart Disease Risk Scale (PHDRS) was developed in 2008 by Ammouri and Neuberger with the objective of determining individuals' perceived risk of developing heart disease. A study was conducted in 2016 by Toptaner and Yıldız to ascertain the scale's validity and reliability in the Turkish population. The scale is composed of 20 items and three sub-dimensions, and utilises a 4-point Likert scale.
Framingham Risk Score | From 01 January 2023 to 01 Februrary 2023 (4 weeks)
  The Framingham Risk Score is a widely used and reliable method of estimating an individual's 10-year risk of developing CHD. The calculation takes into account six risk factors: gender, age, LDL cholesterol, HDL cholesterol, diabetes, blood pressure and smoking status. Based on these values and categories, scores are determined and the corresponding 10-year risk probability is calculated. A score of less than 10% indicates low risk, 10-20% indicates moderate risk, and more than 20% indicates high risk.

SECONDARY OUTCOMES:
Knowledge Level of Cardiovascular Disease Risk Factors Scale | From 15 June 2023 to 15 July 2023 (4 weeks)
  The Knowledge Level of Cardiovascular Disease Risk Factors Scale (KL-CDRFS) was developed and validated by Arıkan et al. in 2009. Notably, it is the inaugural scale in Turkey to have been both validated and proven reliable for the purpose of assessing knowledge levels concerning cardiovascular disease risk factors (Cronbach's alpha: 0.768). The scale comprises 28 items, and evaluation is based on the total score obtained. Participants respond to items with "Yes," "No," or "I don't know," and correct responses are scored as 1 point. It is important to note that, in the interest of scientific rigour, any responses marked as "I don't know" are categorised as incorrect during the evaluation process, thus ensuring the integrity of the data collected.
Perception of Heart Disease Risk Scale | From 15 June 2023 to 15 July 2023 (4 weeks)
  The Perception of Heart Disease Risk Scale (PHDRS) was developed in 2008 by Ammouri and Neuberger with the objective of determining individuals' perceived risk of developing heart disease. A study was conducted in 2016 by Toptaner and Yıldız to ascertain the scale's validity and reliability in the Turkish population. The scale is composed of 20 items and three sub-dimensions, and utilises a 4-point Likert scale.
Framingham Risk Score | From 15 June 2023 to 15 July 2023 (4 weeks)
  The Framingham Risk Score is a widely used and reliable method of estimating an individual's 10-year risk of developing CHD. The calculation takes into account six risk factors: gender, age, LDL cholesterol, HDL cholesterol, diabetes, blood pressure and smoking status. Based on these values and categories, scores are determined and the corresponding 10-year risk probability is calculated. A score of less than 10% indicates low risk, 10-20% indicates moderate risk, and more than 20% indicates high risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Dursun Odabaş Medicine Center, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No